CLINICAL TRIAL: NCT01039285
Title: Exogenous Surfactant in Very Preterm Neonates Presenting With Severe Respiratory Distress in Prevention of Bronchopulmonary Dysplasia
Brief Title: Exogenous Surfactant in Very Preterm Neonates in Prevention of Bronchopulmonary Dysplasia
Acronym: CURDYS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jean Michel Hascoet (Other)
Collaborators: ARAIRLOR (Unknown); Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor-Investigator, Jean Michel Hascoet, Professor, Maternite Regionale Universitaire
Organization: Maternite Regionale Universitaire (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRU-09-02; 2009-012817-23 (Registry Identifier: EUDRACT)
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Infant, Premature, Diseases; Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia
Keywords: Very premature infant; Surfactant; Respiratory Distress; Bronchopulmonary Dysplasia
MeSH Terms: conditions — Infant, Premature, Diseases; Respiratory Distress Syndrome, Newborn; Bronchopulmonary Dysplasia; Dyspnea | interventions — poractant alfa; Air

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surfactant instillation (Experimental): 2.5 ml/kg of Surfactant will be instilled in the trachea
  Interventions: Drug: Curosurf
- Placebo instillation (Placebo Comparator): 2.5 ml/kg of Air will be instilled in the trachea
  Interventions: Other: Air

INTERVENTIONS:
Drug: Curosurf — 2.5 ml/kg instilled in the trachea
  Arms: Surfactant instillation
Other: Air — 2.5ml/kg of Air will be instilled in the trachea
  Arms: Placebo instillation

SUMMARY:
Advances in perinatal care have made it possible to improve the survival of the most immature neonates, but at the cost of an increase in the population at risk of developing bronchopulmonary dysplasia (BPD). Measures that have attempted to limit the development of BPD are not always effective, or related to major side effects. The physiopathological factors that are identified in BPD should, in theory, respond to surfactant. Therefore, the use of an exogenous surfactant in neonates presenting with pulmonary disease requiring mechanical ventilation, leading to a significant risk of BPD, should allow earlier extubation and thus promote pulmonary healing and growth.

ELIGIBILITY:
Inclusion Criteria:

* any neonate of gestational age less than 33 weeks of amenorrhea still on conventional assisted ventilation or HFOV (High Frequency Oscillatory Ventilation), after 14 ± 2 days of life

Exclusion Criteria:

* active infection (CRP > 30 mg/L) not controlled by appropriate antibiotic treatment
* use of corticosteroids in the postnatal period
* significant neurological or malformative disease
* surgical intervention < 72 hours
* refusal of parental approval

Ages: 12 Days to 16 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 118 (Actual)
Dates: Start 2009-12 (Actual); Primary Completion 2021-09 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
duration of assisted ventilation | days
  we aim to demonstrate a significant reduction in the duration of assisted ventilation in children presenting with severe respiratory distress at 14+/-2 days of life.

SECONDARY OUTCOMES:
to reduce the incidence of BPD | 36 weeks post conceptional age
to improve the inflammatory status of the lung and to restore its capacities for healing and growth | one month
to improve development in stature and weight, psychomotor development, and to reduce respiratory sequelae leading to re-hospitalisation | 2 years of age
to improve height development, psychomotor development and respiratory function | 7 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel HASCOET, MD, Study Director — Maternite Regionale Universitaire NANCY
Locations (13):
- France (13):
  - CHU Hopital Nord, Amiens
  - CHU, Angers
  - Centre Hospitalier, Arras
  - CHU Hopital Clemenceau, Caen
  - CHU hopital d'enfants, Dijon
  - Centre Hospitalier, Lens
  - CHU Hopital Jeanne de Flandre, Lille
  - CHU Hopital de la Croix Rousse, Lyon
  - APHM hopital de la conception, Marseille
  - CHI Andre Gregoire, Montreuil
  - Maternite Regionale Universitaire, Nancy
  - AP-HP Hopital Port Royal, Paris
  - CHU Hopital Gatien de Clocheville, Tours

REFERENCES:
- [Result] Hascoet JM, Picaud JC, Ligi I, Blanc T, Moreau F, Pinturier MF, Zupan V, Guilhoto I, Hamon IR, Alexandre C, Bouissou A, Storme L, Patkai J, Pomedio M, Rouabah M, Coletto L, Vieux R. Late Surfactant Administration in Very Preterm Neonates With Prolonged Respiratory Distress and Pulmonary Outcome at 1 Year of Age: A Randomized Clinical Trial. JAMA Pediatr. 2016 Apr;170(4):365-72. doi: 10.1001/jamapediatrics.2015.4617. PMID 26928567
- [Result] Hascoet JM, Picaud JC, Ligi I, Blanc T, Daoud P, Zupan V, Moreau F, Guilhoto I, Rouabah M, Alexandre C, Saliba E, Storme L, Patkai J, Pomedio M, Hamon I. Review shows that using surfactant a number of times or as a vehicle for budesonide may reduce the risk of bronchopulmonary dysplasia. Acta Paediatr. 2018 Jul;107(7):1140-1144. doi: 10.1111/apa.14171. Epub 2017 Dec 22. PMID 29193276